CLINICAL TRIAL: NCT03625297
Title: Shelter Cat Adoption in Families of Children With Autism: Impact on Cat Stress and Children's Social Skills and Anxiety ("Feline Friends")
Brief Title: Shelter Cat Adoption in Families of Children With Autism (Feline Friends)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Winn Feline Foundation (Unknown); Human Animal Bond Research Institute (HABRI) (Unknown)
Responsible Party: Principal Investigator, Gretchen K Carlisle, Research Scientist, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2008460
Record Dates: First submitted 2018-07-17; First posted 2018-08-10 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Social Skills; Anxiety
MeSH Terms: conditions — Social Skills; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study uses a two-group randomized, repeated measures design with a delayed treatment control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shelter cat adoption control group (No Intervention): Families of children with autism will complete a control period with no intervention, then adopt a shelter cat after completion of the control period
- shelter cat adoption (Experimental): Families of children with autism will adopt a shelter cat
  Interventions: Other: shelter cat

INTERVENTIONS:
Other: shelter cat — families will adopt a shelter cat
  Arms: shelter cat adoption

SUMMARY:
The overall purpose of this study is to investigate the effect of the introduction of a shelter cat into the family of a child with Autism Spectrum Disorder on the social skills and anxiety of the child, and to examine stress in the cat.

DETAILED DESCRIPTION:
Many families in the United States live with cats as companion animals, including families of children with Autism Spectrum Disorder (ASD). One in 68 children are diagnosed with ASD. There is no cure for ASD, and no one treatment works for all children. Symptoms of ASD include a lack of social skills and anxiety. Companion animals have been helpful for children with ASD. However, no one has studied stress of cats living in families of children with ASD. This study will place 64 pre-screened shelter cats in pre-screened homes and monitor the stress of the cats. Cats ages 10 months to four years that have been screened for calm behavior using a temperament, test will be adopted by families in the study. Families will also be screened for pet issues. No cat will be placed in a home with a child who has a history of aggression to animals. The study will also examine the social skills and anxiety of the children with ASD, and bonding of the parents and children with their cats. Five to eight million dogs and cats are relinquished to animal shelters in the United States each year. Thirty-eight percent of cats are given up for behavioral reasons. Studying cat stress and the placement of cats, with calm and non-aggressive characteristics into homes of families of children with ASD may help shed light on the likely success of the relationships between shelter cats and these families.

ELIGIBILITY:
Inclusion Criteria:

* child with diagnosis of Autism Spectrum Disorder
* no cat currently living with the family
* willingness to adopt a shelter cat
* English speaking
* live within 125 miles of Columbia, Missouri

Exclusion Criteria:

* child with Autism Spectrum Disorder having any history of animal aggression
* children with cat allergies

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Social Skills of child with autism over time from baseline to 6, to 12 and to 18 weeks | Control: Baseline, 6, 12 and 18 weeks Treatment: Baseline, 6, 12 and 18 weeks
  Social skills measured using the Social Skills Improvement System Rating Scale (SSiS-RS) with scores from 0-138.
Change in Anxiety of child with autism over time from baseline to 6, to 12 and to 18 weeks | Control: Baseline, 6, 12 and 18 weeks Treatment: Baseline, 6, 12 and 18 weeks
  Anxiety measured using the Screen for Child Related Anxiety Disorders (SCARED) with scores from 0-82.

SECONDARY OUTCOMES:
change in parent Human-animal Bonding over time from 2-3 days, to 6, to 12 and 18 weeks | Baseline, 6, 12 and 18 weeks Treatment: Baseline, 2-3 days, 6, 12 and 18 weeks
  bonding of parent and cat using Lexington Attachment to Pets Scale with scores from 0-54.
change in child Human-animal Bonding over time from 2-3 days, to 6, to 12 and 18 weeks | Baseline, 6, 12 and 18 weeks Treatment: Baseline, 2-3 days, 6, 12 and 18 weeks
  bonding of child with autism and cat using the Companion Animal Bonding Scale with scores from 8-40

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen K Carlisle, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States